CLINICAL TRIAL: NCT05867069
Title: Knee MRI and Markerless Motion Capture Analysis in Patients With Femoroacetabular Impingement Syndrome
Brief Title: Analysis of Radiographic and Kinematic Features in FAI Patients
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S2021436
Record Dates: First submitted 2023-04-25; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Femoro Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ipsilateral knee pain group: Those FAI patients presenting with preoperative ipsilateral knee pain.
- No ipsilateral knee pain group: Those FAI patients presenting without preoperative ipsilateral knee pain.

SUMMARY:
The goal of this observational study is to describe the radiographic and kinematic features in patients with femoroacetabular impingement syndrome (FAI). The main questions it aims to answer are:

* Is structural knee abnormalities associated with knee pain symptoms in FAI patients?
* Does FAI patients with knee pain demonstrate unique kinematic characteristics？ Participants will receive routine preoperative radiographic examinations, which include ipsilateral knee MRI for the purpose of femoral version measurement. Participants will also receive markerless motion capture analysis.

Researchers will compare preoperative radiographic and kinematic features based on knee pain status, which is routinely collected as part of clinical investigation procedures.

DETAILED DESCRIPTION:
This observational study aims to study the association between preoperative subjective knee pain and baseline knee radiographic and kinematic characteristics. MRI of the ipsilateral knee is screened for structural abnormalities, including cartilage defects, meniscal tears and ligament injuries. Markerless motion capture data are evaluated for transverse plane kinematic features, with a primary focus on foot progression angles during normal gait.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed with FAI based on clinical and radiographical findings;
* (2) failed conservative treatment for at least 6 months and indicated for surgical treatment;
* (3) received routine preoperative hip and ipsilateral knee MRI.

Exclusion Criteria:

* (1) history of fracture or surgery of hip and knee;
* (2) avascular necrosis;
* (3) Legg-Calve-Perthes disease;
* (4) Ehlers-Danlos syndrome;
* (5) pigmented villonodular synovitis (PVNS);
* (6) osteoid osteoma (OO);
* (7) synovial chondromatosis;
* (8) severe hip osteoarthritis (OA) with Tönnis grade > 1;
* (9) developmental dysplasia of hip (DDH)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients diagnosed with FAI and admitted into the sports medicine department at Peking university third hospital for hip arthroscopic surgery by a single surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Preoperative radiographic cartilage defect of ipsilateral knee | Knee MRI radiographs are evaluated at baseline.
  On the same day of admission, patients receive routine preoperative MRI examination of the hip and ipsilateral knee for femoral version measurement. Radiographs of ipsilateral knee MRI are evaluated for the presence of structural knee abnormality. Radiographic signs suggesting cartilage defect of the patella, femur and the tibial plateau are collected.
Preoperative radiographic meniscal tear of ipsilateral knee | Knee MRI radiographs are evaluated at baseline.
  On the same day of admission, patients receive routine preoperative MRI examination of the hip and ipsilateral knee for femoral version measurement. Radiographs of ipsilateral knee MRI are evaluated for the presence of structural knee abnormality. Radiographic signs suggesting lateral or medial meniscal tears are collected.
Preoperative radiographic ligament ruptures of ipsilateral knee | Knee MRI radiographs are evaluated at baseline.
  On the same day of admission, patients receive routine preoperative MRI examination of the hip and ipsilateral knee for femoral version measurement. Radiographs of ipsilateral knee MRI are evaluated for the presence of structural knee abnormality. Radiographic signs suggesting ACL tears, PCL tears or collateral ligament ruptures are collected.
Foot progression angle during normal gait | Motion capture data are assessed at baseline.
  The next day after admission, patients undergo markerless motion capture evaluation after informed consents are obtained. Movements for motion capture include normal gait, stepping in place, single-leg stance, double-leg squat and forward lunge. Each movement is repeated 2 times. The entire data collection process for each patient takes approximately 120 seconds. Foot progression angle during gait are assessed with MATLAB in a retrospective fashion after completion of patient recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xu, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No